CLINICAL TRIAL: NCT07389928
Title: Comprehensive Biomarker ProfiliNg in PatieNts With VEntriCular TachyCardia, PremAtuRe VEntricular Contractions, and AVNRT (CONNECT-CARE)
Brief Title: Comprehensive Biomarker ProfiliNg in PatieNts With VEntriCular TachyCardia, PremAtuRe VEntricular Contractions, and AVNRT
Acronym: CONNECT-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Roland Richard Tilz, MD, Director, Department of Rhythmology, University of Luebeck
Other Study IDs: CONNECT-CARE
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General cohort

SUMMARY:
To systematically evaluate multiple biomarkers in patients ventricular tachycardia (VT), premature ventricular contractions (PVC), atrioventricular nodal reentrant tachycardia (AVNRT) undergoing catheter ablation to elucidate their mechanistic relevance and predictive value.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Catheter ablation due to VT, PVC, or AVNRT
* Written informed consent

Exclusion criteria:

* Infection or inflammatory disease at time of sampling
* Pregnancy
* Inability to comply with study procedures
* Life expectancy < 1 year not due to arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ventricular tachycardia (VT), premature ventricular contractions (PVC), atrioventricular nodal reentrant tachycardia (AVNRT) undergoing catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Association between baseline biomarker profiles and arrhythmia subtype (VT, PVC, AVNRT). | 24 months

IPD SHARING:
Plan to Share IPD: Undecided